CLINICAL TRIAL: NCT02757053
Title: Screening Brain MRI in High School Football: What is the Risk of Traumatic Brain Injury and Does the Guardian Cap Reduce the Incidence of Injury as Determined by Fluid-attenuated Inversion Recovery (FLAIR) and Susceptibility Weighted Imaging (SWI) Magnetic Resonance Imaging (MRI) Sequences
Brief Title: Screening Brain MRI in High School Football: Does the Guardian Cap Reduce the Risk of Traumatic Brain Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was terminated June 28 2016 for low enrollment and PI moving away. No results were obtained
Sponsor: Mosaic Life Care (Other)
Collaborators: Missouri Western State University (Unknown)
Responsible Party: Principal Investigator, Paul Isenbarger, Diagnostic and Interventional Radiologist, Mosaic Life Care
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MLC002
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2016-08

CONDITIONS: Brain Concussion; Brain Injuries; Diffuse Axonal Injury; Athletic Injuries; Injury, Brain, Traumatic
Keywords: Brain Concussion; Brain Injuries; Diffuse Axonal Injury; Football; Head Protective Devices; Magnetic Resonance Imaging; Helmet; Third party add-on
MeSH Terms: conditions — Brain Concussion; Brain Injuries; Diffuse Axonal Injury; Athletic Injuries; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guardian Cap (Experimental): The set of high school football players wearing the Guardian Cap on their helmets
  Interventions: Device: Guardian Cap
- No Guardian Cap (No Intervention): The set of high school football players not wearing the Guardian Cap on their helmets

INTERVENTIONS:
Device: Guardian Cap — The Guardian Cap is a third party add-on device attached to the facemask of a football helmet that covers the outside of the helmet with a soft material to reduce the initial impact severity, thus reducing the forces transmitted to the brain
  Other Names: Third party add-on
  Arms: Guardian Cap

SUMMARY:
Screening Brain magnetic resonance imaging (MRI) with Fluid-attenuated Inversion Recovery (FLAIR) and Susceptibility Weighted Imaging (SWI) sequences will be performed pre and post season on high school football players. One set of players will wear the Guardian Cap on their five star rated helmets and the other will wear five star rated helmets only. The investigators will compare outcomes of ImPACT scores and MRI findings between the two groups to see if there is a statistical difference in reduction of injury and to establish what the baseline level of MRI findings related to injury from high school football is as well as what the baseline level of injury is prior to the start of the season.

DETAILED DESCRIPTION:
Screening Brain Magnetic Resonance Imaging (MRI) with Fluid-attenuated Inversion Recovery (FLAIR) and Susceptibility Weighted Imaging (SWI) sequences will be performed pre and post season on high school football players. One set of players will wear the Guardian Cap on their five star rated helmets and the other will wear five star rated helmets only. The investigators will compare outcomes of ImPACT concussion scores and MRI findings on FLAIR and SWI sequences between the two groups to see if there is a statistical difference in reduction of MRI findings on FLAIR and SWI sequences or adverse ImPACT concussion score outcomes and to establish what the baseline level of MRI findings on FLAIR and SWI sequences related to injury from high school football is as well as what the baseline level of MRI findings on FLAIR and SWI is prior to the start of the season.

ELIGIBILITY:
Inclusion Criteria:

* High school football players willing and able to have a pre and post season Brain MRI with FLAIR and SWI sequences and wear the Guardian Cap on their helmet

Exclusion Criteria:

* High school football players unwilling or unable to have an MRI

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06-14 (Actual); Study Completion 2016-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Isenbarger, MD, Principal Investigator — Daignostic and Interventional Radiologist at Mosaic Life care
Locations (1):
- Mosaic Life Care, Saint Joseph, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share data with MRI results of individual exams with the patient and plan to publish in peer reviewed journal

REFERENCES:
- [Background] Beauchamp MH, Beare R, Ditchfield M, Coleman L, Babl FE, Kean M, Crossley L, Catroppa C, Yeates KO, Anderson V. Susceptibility weighted imaging and its relationship to outcome after pediatric traumatic brain injury. Cortex. 2013 Feb;49(2):591-8. doi: 10.1016/j.cortex.2012.08.015. Epub 2012 Sep 3. PMID 23062584
- [Background] Mittl RL, Grossman RI, Hiehle JF, Hurst RW, Kauder DR, Gennarelli TA, Alburger GW. Prevalence of MR evidence of diffuse axonal injury in patients with mild head injury and normal head CT findings. AJNR Am J Neuroradiol. 1994 Sep;15(8):1583-9. PMID 7985582

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was prematurely terminated due to the PI leaving the area. A few participants did enroll with baseline data only being collected prior to termination.
Period: Overall Study
Arm/Group | Guardian Cap | No Guardian Cap
Started | 3 | 5
Completed | 0 | 0
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guardian Cap | No Guardian Cap | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 5 | 8
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: MRI Brain SWI and FLAIR Lesions Pre and Post High School Football Season With and Without the Guardian Cap
Description: MRI Brain SWI Lesions pre and post football season with and without the Guardian Cap
Time Frame: within the first two months after the high school football season ends
Population: Study was prematurely terminated due to the PI leaving the area. A few participants did enroll with baseline data only being collected prior to termination. No outcome data collected.
Arm/Group | Guardian Cap | No Guardian Cap
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: ImPact Concussion Scores Pre and Post High School Football Season With and Without the Guardian Cap
Description: Establish the expected range of ImPact concussion scores pre and post football season with and without the Guardian Cap
Time Frame: within the first two months after the high school football season ends
Population: as for outcome 1
Arm/Group | Guardian Cap | No Guardian Cap
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of MRI Brain SWI and FLAIR Lesions in Preseason High School Football Players
Description: Establish the expected range of MRI Brain SWI and FLAIR lesions in the general high school population at the beginning of a high school football season
Time Frame: within two months of the start of high school football season
Population: as for outcome 1
Arm/Group | Guardian Cap | No Guardian Cap
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of MRI Brain SWI and FLAIR Lesions in Postseason High School Football Players
Description: Establish the incidence of MRI Brain SWI and FLAIR lesions in postseason high school football players
Time Frame: within two months of the end of high school football season
Population: as for outcome 1
Arm/Group | Guardian Cap | No Guardian Cap
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Study was prematurely terminated due to the PI leaving the area. A few participants did enroll with baseline data only being collected prior to termination. No adverse event information collected.
Arm/Group | Guardian Cap | No Guardian Cap
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No